CLINICAL TRIAL: NCT07385963
Title: EIT-Based Pulmonary Perfusion Pulse Wave Versus Swan-Ganz Catheter in Stroke Volume Correlation
Brief Title: Correlation Between EIT-based Pulse Wave Method for Pulmonary Perfusion Monitoring and Pulmonary Artery Catheter-based Stroke Volume Measurement
Acronym: EIT-Cath Corre
Status: Not yet recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: EITSV20240717; EITSV20240717 (Other: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology)
Record Dates: First submitted 2025-12-11; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Shock; Acute Respiratory Distress Syndrome
Keywords: Critical Illness; Acute Respiratory Distress Syndrome; Shock; Hemodynamic Monitoring; Electric Impedance; Pulmonary Circulation
MeSH Terms: conditions — Shock; Respiratory Distress Syndrome; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples Without DNA — EIT Images and Signal Data: Dynamically sequenced lung perfusion images and raw impedance waveforms collected by the electrical impedance tomography device.
  Hemodynamic Data: Measurements from the Swan-Ganz catheter synchronized with EIT monitoring, including parameters such as stroke volume.
  Respiratory Mechanics Data: Parameters recorded during mechanical ventilation, including airway pressure, tidal volume, and PEEP settings.
  Anonymized Clinical Data: De-identified basic clinical information of patients corresponding to the data mentioned above.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Catheter Cohort: This cohort enrolls all critically ill patients who meet the inclusion criteria, including those requiring mechanical ventilation, meeting the 2023 global ARDS definition and/or being in shock requiring vasoactive drugs, and who have already had a Swan-Ganz catheter inserted for clinical reasons. This study is observational in design and does not impose any additional therapeutic interventions. During the study period, the pulmonary perfusion signals measured by the Electrical Impedance Tomography (EIT) pulse wave method and the actual cardiac stroke volume (SV) data measured by the Swan-Ganz catheter will be recorded synchronously and compared to analyze their correlation and establish a regression model. All monitoring is part of routine medical care based on the patient's clinical condition.
  Interventions: Diagnostic Test: Synchronous Data Acquisition of EIT and Pulmonary Artery Catheter

INTERVENTIONS:
Diagnostic Test: Synchronous Data Acquisition of EIT and Pulmonary Artery Catheter — This study is observational in design and does not impose any therapeutic interventions. The described "intervention" refers to the synchronous data acquisition process performed for research purposes. Specifically, based on routine clinical monitoring, the timing of EIT pulse wave method for pulmonary perfusion monitoring and Swan-Ganz catheter for stroke volume (SV) monitoring is precisely synchronized (to the second), and data from both are recorded for subsequent correlation and regression analysis. All monitoring methods are required for the patient's clinical diagnosis and treatment; the research activity is limited to the synchronous recording and comparison of data.
  Other Names: This field does not need to be filled as there are no other defined interventions in the study.

SUMMARY:
The goal of this clinical study is to learn if a new, non-invasive monitoring method called EIT Pulse Wave can accurately measure blood flow to the lungs (pulmonary perfusion) and predict heart stroke volume (SV) in critically ill patients. It will also learn about the safety of this monitoring approach. The main questions it aims to answer are:

How well does the EIT Pulse Wave measurement of lung blood flow correlate with the SV measured by the standard method (Swan-Ganz catheter)? Can we build a reliable model to predict SV non-invasively using the EIT Pulse Wave signal? Researchers will compare the EIT Pulse Wave measurements directly with the Swan-Ganz catheter measurements to see if the new method is accurate.

Participants will:

Be critically ill adults in the ICU who are already receiving mechanical ventilation and have a Swan-Ganz catheter in place for medical reasons.

Undergo simultaneous monitoring using both the EIT device and the Swan-Ganz catheter every 30 minutes for up to 48 hours.

Have their ventilator settings adjusted to different levels as part of the study protocol while both measurements are recorded.

DETAILED DESCRIPTION:
Research Overview: Developing a Safer and Simpler Method to Monitor Heart and Lung Function in Critically Ill Patients

1. Why are we conducting this study? In the intensive care unit (ICU), doctors need to constantly track subtle changes in patients' heart and lung function, particularly how much blood the heart pumps with each beat (known as "stroke volume") and how blood flows through the lungs (known as "pulmonary perfusion"). This information is crucial for precise medication administration and adjusting ventilator settings.

   Currently, the "gold standard" method for measuring stroke volume requires inserting a long, thin catheter (a Swan-Ganz catheter) into a patient's major blood vessel, advancing it near the heart. This is an invasive procedure that carries risks such as infection and bleeding, is expensive, and is technically complex.

   Therefore, there is an urgent need to find a non-invasive, safe, and simple method that can continuously and in real-time monitor these critical indicators, much like tracking heart rate or blood pressure.
2. What new method are we testing? We are studying a brand-new technology called "Electrical Impedance Tomography (EIT) Pulse Wave Method." You can think of it as a "smart camera," but instead of using radiation, it uses very weak, safe electrical currents-imperceptible to the human body-to "see" blood flow in the lungs.

   The advantages of this technology are significant:

   Completely Non-Invasive: It only requires placing a belt with electrodes on the patient's chest, causing no trauma.

   Real-Time Bedside Monitoring: The device can be brought to the bedside, providing continuous, dynamic images and data without moving critically ill patients.

   Radiation-Free: It poses no risk of radiation exposure to either patients or medical staff.
3. What is the core question this study aims to answer? While the EIT Pulse Wave method is technologically advanced, we do not yet know if the "pulmonary perfusion signal" it measures is accurate and reliable. Can the data it captures truly reflect the volume of blood pumped by the heart? This is the goal of our study: to conduct a head-to-head, precise comparison between this new non-invasive method and the traditional invasive "gold standard" method to verify its reliability.
4. How will the study be conducted? Study Type: This is an observational study. This means we will not make any additional interventions to the patient's treatment. We will only simultaneously record data measured by both devices at the same time points.

   Participants: We will recruit critically ill patients who require a Swan-Ganz catheter for their own medical condition. Their participation will not introduce additional medical risks.

   Research Process: After patients consent to join the study, we will initiate the non-invasive EIT monitoring simultaneously with the routine stroke volume measurements taken via the Swan-Ganz catheter. We will pair and compare the data recorded by both devices at identical time points (accurate to the second).
5. What potential benefits might this study bring? For Future Patients: If the study is successful and proves the EIT Pulse Wave method is reliable, countless future critically ill patients could benefit. They could avoid the pain and risks associated with invasive catheters while receiving more continuous and convenient monitoring of heart and lung function, leading to more precise, individualized treatment.

For Medical Progress: This would introduce a revolutionary tool to the field of critical care medicine, advancing the development of "non-invasive monitoring" technologies, and ultimately potentially reducing healthcare costs and improving patient outcomes.

For the Participants Themselves: While participation in this study may not offer direct therapeutic benefits, the intensive data monitoring might provide the medical team with richer physiological information, potentially helping to optimize their current treatment plan.

In summary, this study aims to take the crucial first step: validating a promising non-invasive technology, with the hope of transforming the monitoring methods for critically ill patients in the future, making treatment safer and more precise.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients requiring mechanical ventilation support.
* Patients meeting the 2023 global ARDS definition and/or shock patients receiving vasoactive medication therapy.
* Patients who have already had a pulmonary artery catheter inserted due to clinical needs.

Exclusion Criteria:

* Age under 18 years or over 80 years.
* Patients with severe obesity (BMI ≥ 35 kg/m²).
* Pregnant or lactating women.
* Pulmonary embolism.
* Patients undergoing ECMO therapy.
* Arrhythmia.
* Contraindications to EIT monitoring.
* Contraindications to pulmonary artery catheter use.
* Failure to provide signed informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of critically ill adult patients admitted to the Intensive Care Unit of Union Hospital, Tongji Medical College, Huazhong University of Science and Technology. All participants require mechanical ventilation support and meet either the 2023 global ARDS diagnostic criteria and/or are receiving vasoactive medications for shock treatment. A key inclusion prerequisite is that patients must already have a Swan-Ganz catheter inserted for clinical hemodynamic monitoring purposes. Study subjects will undergo simultaneous non-invasive EIT monitoring and invasive catheter measurements to evaluate the correlation between the two methods in measuring stroke volume.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between EIT Pulmonary Perfusion Signal and Catheter-measured Stroke Volume | From the start of synchronous monitoring for each enrolled subject until the end of the monitoring period (up to 48 hours).
  Outcome Measure Title: EIT-derived stroke perfusion signal value, measured via the pulse wave analysis method of Electrical Impedance Tomography (EIT) equipment.
  Measuring Tool: Electrical Impedance Tomography (EIT) system and its accompanying pulse wave analysis software.
  Unit of Measure: Relative impedance change units (or Arbitrary Units). Time Point Description: Recorded at each time point synchronized with pulmonary artery catheter measurements, starting from study inclusion, every 30 minutes, for a maximum duration of 48 hours.
  Primary Outcome Measure 2: Cardiac Stroke Volume Measured by Pulmonary Artery Floating Catheter
  Outcome Measure Title: Stroke volume, measured via continuous cardiac output monitoring using a pulmonary artery floating catheter (Swan-Ganz catheter).
  Measuring Tool: Pulmonary artery floating catheter and its accompanying cardiac output monitor.
  Unit of Measure: Milliliters per beat (mL/beat). Time Point Description: Recorded

SECONDARY OUTCOMES:
Correlation of HPB (EIT) and CO (Swan-Ganz catheter) | at the time of 48 hours after inclusion.
  Continuous monitoring of patients' HPB values was performed using an EIT device, while cardiac output (CO) was simultaneously measured using a Swan-Ganz catheter. Depending on the distribution of the data (normal or non-normal), Pearson or Spearman correlation analysis was applied to calculate the correlation coefficient and the corresponding P value between HPB and CO.
Correlation of HPB (EIT) and SV (Swan-Ganz catheter) | at the time of 48 hours after inclusion
  Continuous monitoring of patients' HPB values was performed using an EIT device, while stroke volume (SV) was simultaneously measured using a Swan-Ganz catheter. Depending on the distribution of the data (normal or non-normal), Pearson or Spearman correlation analysis was applied to calculate the correlation coefficient and the corresponding P value between HPB and SV.
Correlation between EISV measured by EIT and cardiac output (CO) measured by Swan-Ganz catheter | at the time of 48 hours after inclusion
  Continuous monitoring of patients' HPB values was performed using an EIT device, while cardiac output (CO) was simultaneously measured using a Swan-Ganz catheter. Depending on the distribution of the data (normal or non-normal), Pearson or Spearman correlation analysis was applied to calculate the correlation coefficient and the corresponding P value between EISV and CO.
Correlation between EISV measured by EIT and stroke volume (SV) measured by Swan-Ganz catheter | at the time of 48 hours after inclusion
  Continuous monitoring of patients' HPB values was performed using an EIT device, while stroke volume (SV) was simultaneously measured using a Swan-Ganz catheter. Depending on the distribution of the data (normal or non-normal), Pearson or Spearman correlation analysis was applied to calculate the correlation coefficient and the corresponding P value between EISV and SV.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be shared due to participant privacy and data protection concerns. The datasets contain detailed clinical information that, even after de-identification, could potentially allow for re-identification of individuals given the specific and critical nature of the patient population. Furthermore, a comprehensive data sharing agreement plan has not been established for this study.

REFERENCES:
- [Result] Fujita Y, Kent M, Wisner E, et al. Combined assessment of pulmonary ventilation and perfusion with single-energy computed tomography and image processing. Acad Radiol,2021, 28:636-646.
- [Result] Nguyen DT, Jin C, Thiagalingam A, et al. A review on electrical impedance tomography for pulmonary perfusion imaging. Physiol Meas, 2012, 33(5): 695-706.
- [Result] Franchineau G, Jonkman AH, Piquilloud L, et al.Electrical Impedance Tomography to Monitor Hypoxemic Respiratory Failure. Am J Respir Crit Care Med.2024.15;209(6):670-682
- [Result] Frerichs I, Amato MBP, Van Kaam AH, et al. Chest electrical impedance tomography examination, data analysis, terminology, clinical use and recommendations:Consensus statement of the translational EIT development study group. Thorax, 2017, 72(1):83-93